CLINICAL TRIAL: NCT00416702
Title: An Open-Label, Single-Dose, Parallel-Group Study to Assess the Pharmacokinetics of 600 µg Indacaterol in Subjects With Impaired Hepatic Function in Comparison With Healthy Control Subjects
Brief Title: Safety and Pharmacokinetics of Indacaterol in Healthy Subjects and Those With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149A2307
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Hepatic Insufficiency
Keywords: safety study, pharmacokinetic effects, healthy subjects, hepatic impairment, liver; Subjects with mild and moderate hepatic impairment and healthy subjects
MeSH Terms: conditions — Hepatic Insufficiency | interventions — indacaterol

ARMS (1):
- 1 (Experimental): QAB149
  Interventions: Drug: QAB149

INTERVENTIONS:
Drug: QAB149
  Other Names: indacaterol

SUMMARY:
This study is designed to evaluate the safety and pharmacokinetic effects of indacaterol in subjects with impaired liver function in comparison with healthy subjects

ELIGIBILITY:
Inclusion Criteria:

All Groups

* Male and/or female subjects in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Female subjects of child bearing potential must be using a double-barrier local contraception, i.e. intra-uterine device plus condom, or spermicidal gel plus condom or oral contraception.
* OR:

Postmenopausal women must have no regular menstrual bleeding for at least 1 years prior to inclusion. Menopause will be confirmed by a plasma FSH level of >40 IU/L

OR:

Female subjects must have been surgically sterilized at least 6 months prior to screening.with supportive clinical documentation.

AND/OR and MDS-specific requirement: If female subjects have male partners who have undergone vasectomy, the vasectomy must have occurred more than 6 month prior to first dosing.

All females must have negative pregnancy test results at screening and baseline.

* Subjects must weigh at least 50 kg and have a body mass index (BMI) between 18 and 40 kg/m2 to participate in this study.
* Platelet count > 50,000 X 109/L at screening and baseline.

Group 1 (healthy controls)

* In good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening; subjects without diseases/conditions.
* Vital signs should be within the following ranges: oral body temperature between 35.0-37.5 °C, systolic blood pressure, 90-<140 mm Hg, diastolic blood pressure, 60-<90 mm Hg, pulse rate, 50 - 100 beats per minute (bpm) When blood pressure and pulse will be taken again after at least 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mm Hg drop in diastolic blood pressure and increase in heart rate (>20 bpm) associated with clinical manifestation of postural hypotension.
* Matched with a hepatic impaired patient on a 1:1 ration using the following criteria.sex, age ± 5 years, weight ± 10 kilograms, and smoking status

Group 2, and 3 (hepatic impairment)

* Physical signs consistent with a clinical diagnosis of liver cirrhosis (i.e., liver firmness to palpation, splenic enlargement, spider angioma, palmar erythema, parotid hypertrophy, testicular atrophy, and gynecomastia).
* Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment.
* Otherwise considered healthy in general as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Vital signs should be within the following ranges: oral body temperature between 35.0-37.5 °C, systolic blood pressure, 90-<140 mm Hg, diastolic blood pressure, 60-<90 mm Hg, pulse rate, 50 - 100 beats per minute (bpm).

Exclusion Criteria:

All Groups

* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to study start.
* Significant illness within the 2 weeks prior to study start.
* A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
* Resting heart rate < 50 bpm
* History of autonomic dysfunction or acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated) or clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis), or a known hypersensitivity to the study drug or drugs similar to the study drug .
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study, including bowel, gastrointestinal, renal, pancreatic, hepatic, hematological, immunological, or neurological disorders

Group 1 (healthy controls)

* Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin. SGPT will have to be strictly within the normal range before inclusion, GGT and alkaline phosphatase must not exceed twice the upper limit of the normal range, and serum bilirubin should not exceed the value of 27 µmol/L (1.6 mg/dL).
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Use of any prescription medication within 1 month prior to dosing.
* Use of over-the-counter medications or vitamins within 14 days prior to dosing.
* Vital signs should be within the following ranges: oral body temperature between 35.0-37.5 °C, systolic blood pressure, 90-<140 mm Hg, diastolic blood pressure, 60-<90 mm Hg, pulse rate, 50 - 100 beats per minute (bpm).
* Blood pressure and pulse will be taken again in a standing position. After at least 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 20 bpm increase in pulse rate associated with clinical manifestation of postural hypotension (Otherwise the subject will be classified as experiencing orthostatic hypotension)

Group 2, 3, 4 (hepatic impairment)

* Clinically significant abnormal findings in physical examination, ECG or laboratory evaluations, not consistent with known clinical disease.
* Symptoms or history of Stage II or worse degree of encephalopathy within 6 months of study entry.
* Clinical evidence of severe ascites.
* History of surgical portosystemic shunt.
* Prothrombin time > 18 seconds.
* Any evidence of progressive liver disease (within the last 4 weeks) as indicated by liver transaminases, alkaline phosphatase, and GGT or a ≥ 50% worsening of serum bilirubin or prothrombin time.
* Evidence of drug or alcohol abuse within the last 6 months as indicated by laboratory assays conducted during screening or baseline evaluations.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-11; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessments of orally inhaled indacaterol will be made for up to 168 hours post dose for healthy subjects and for up to 240 hours post dose for patients with mild to moderate liver impairment.

SECONDARY OUTCOMES:
General tolerability and safety indacaterol administered by oral inhalation in the study groups. Safety assessments will include physical examinations, ECGs, vital signs, adverse events, and laboratory evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States